CLINICAL TRIAL: NCT04202926
Title: Repetitive dTMS Intervention for Methamphetamine Addiction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shanghai Mental Health Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: TFYuan
Record Dates: First submitted 2019-11-30; First posted 2019-12-18 (Actual); Last update posted 2023-11-22 (Actual); Status verified 2023-11

CONDITIONS: Methamphetamine-dependence
Keywords: deep transcranial magnetic stimulation; methamphetamine addiction

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 10hz group (Experimental): a high frequency stimulation
  Interventions: Device: real coil
- sham group (Sham Comparator): a sham coil which frequency is 10hz but do not induce stimulation
  Interventions: Device: sham coil

INTERVENTIONS:
Device: real coil — active 10Hz with a train of 3s on / 17s off, 50 trains, a total of 1500 pulses
  Arms: 10hz group
Device: sham coil — sham 10Hz with a train of 3s on / 17s off, 50 trains, a total of 1500 pulses
  Arms: sham group

SUMMARY:
A growing body of evidence suggests a wide range of brain areas including medial prefrontal cortex (mPFC), dorsolateral prefrontal cortex (DLPFC) and other subcortical regions, such as anterior cingulate cortex (ACC) are critical for regulating cognitive control over decisions and involving in drug related cue processing. Previous studies have demonstrated that transcranial magnetic stimulation (rTMS) over dorsolateral prefrontal cortex reduces craving for meth dependences. Specifically, the H7 coil induces a magnetic field can target mPFC and ACC. In this study, the investigators investigated whether repeated dTMS intervention of medial prefrontal and cingulate cortices in methamphetamine addiction could reduce the subjective craving and improve the cognitive abilities.

DETAILED DESCRIPTION:
The study will be conducted at the drug rehabilitation center in China. The whole procedure includes enrollment, pre-intervention evaluation, intervention (for 3 weeks, 5 times a week, 15 times in total), post-intervention evaluation and one month follow up evaluation.

In enrollment session, participants are recruited according to inclusion criteria.

In the pre-intervention evaluation, firstly, participants need complete a questionnaire to assess their demographic information, drug addiction history and drug abstinence. And then are assigned to either 10Hz group or sham group according to the counterbalance of their basic demographic and drug use information. Then, participants need complete craving, cognitive ability and electroencephalogram (EEG) assessment. For craving assessing, participants are shown a video of methamphetamine usage for 5 minutes, and then rated on the visual analogue scale (0 means completely undesired and 100 means extremely wanting) to report their craving for methamphetamine. For cognitive ability and EEG signal assessing, the whole process is conducted on the computer according to instructions.

In the intervention session, dTMS was administered using a TMS stimulator (Magstim, U.K.) equipped with a unique H-shaped coil design. The H-coil version used in this study was the H7 (Brainsway, Jerusalem, Israel). When placed 4-5 cm anterior to the foot motor cortex and used at 100% of the leg resting motor threshold (RMT), the H7 coil stimulates the dorsal mPFC and ACC bilaterally. A participant's RMT was determined before the first treatment and at the beginning of each week by ascertaining the coil position that elicited the minimal involuntary contractions of the feet (three of six attempts). The 10Hz group received 10 Hz dTMS at 100% of RMT, with 3-second pulse and 17-second intervals, for a total of 50 trains and 1500 pulses per session. The sham group received treatment with identical technical parameters, which induced scalp sensations but without penetration of the electric field into the brain.

Post-intervention evaluation and one month follow up evaluation are the same as in pre-intervention evaluation.

To ensure study quality, some measures are taken as bellow:

Researchers and drug rehabilitation staff will work together in whole process and the data will be converted into electronic versions once finishing each evaluation.

In the intervention, patients, operators, and raters were blind to treatment condition. Each patient is assigned a magnetic card that determined the coil (real or sham) in the helmet and raters are not present while treatments are administered.

After each treatment times, any side effect from participant's report are recorded to assure the safety and feasibility.

Statistical analyses are performed using SPSS 21.0. The principal statistical analysis is performed using repeated-measures analysis of variance and regression analysis. All missing data will be recorded and marked.

ELIGIBILITY:
Inclusion Criteria:

* Methamphetamine dependents
* middle school degree or above

Exclusion Criteria:

* Have contraindications to rTMS (head trauma, epilepsy or history of epilepsy, metal implant etc.)
* psychiatric illnesses
* intellectual impairment (IQ<90)

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 23 (Actual)
Dates: Start 2019-12-30 (Actual); Primary Completion 2023-05-30 (Actual); Study Completion 2023-10-30 (Actual)

PRIMARY OUTCOMES:
Changes of Cue-induced craving and ERP | the day before intervention, 3 weeks after intervention, 1 month after intervention, up to 3 months after intervention
  Subjective craving (cue induced, 0-100 based VAS, craving scale) and drug cue-ERP (P300 etc. measured)

SECONDARY OUTCOMES:
Changes of cognition: behavioral inhibition | the day before intervention, 3 weeks after intervention, 1 month after intervention, up to 3 months after intervention
  using cognitive tasks: stop-signal task
Changes of cognition: working memory | the day before intervention, 3 weeks after intervention, 1 month after intervention, up to 3 months after intervention
  using cognitive tasks: n-back task
Changes of depression status | the day before intervention, 3 weeks after intervention, 1 month after intervention, up to 3 months after intervention
  depression (Beck Depression inventory scale), high score means worse depression
Changes of anxiety status | the day before intervention, 3 weeks after intervention, 1 month after intervention, up to 3 months after intervention
  Anxiety (Beck anxiety inventory scale), higher score means worse anxiety
Changes of sleep status | the day before intervention, 3 weeks after intervention, 1 month after intervention, up to 3 months after intervention
  sleep status measurements (Pittsburgh Sleep Quality Index scale), higher score means worse sleep
Changes of impulsivity | the day before intervention, 3 weeks after intervention, 1 month after intervention, up to 3 months after intervention
  Impulsivity scale (The Barratt Impulsiveness Scale), higher score means higher impulsivity
Changes of resting EEG network | the day before intervention, 3 weeks after intervention, 1 month after intervention, up to 3 months after intervention
  resting EEG signal (Alpha, Beta, Theta, etc) measurement with 128 Channel EGI system

OTHER OUTCOMES:
side effect measurements | every day after each intervention time for the 3 weeks intervention time period
  Side effect scale, including headache, pricking, sleeplessness etc.

CONTACTS AND LOCATIONS:
Overall Officials: Tifei Yuan, PhD, Principal Investigator — Shanghai Mental Health Center
Locations (1):
- Nanjing Dalianshan Addiction Rehab Center, Nanjing, China

IPD SHARING:
Plan to Share IPD: Yes
share all IPD that underlie results in a publication
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Within twelve months after the trial complete
Access Criteria: share to health care personnel, patients and the general public.
URL: http://clinicaltrials.gov

REFERENCES:
- [Background] Shen Y, Cao X, Tan T, Shan C, Wang Y, Pan J, He H, Yuan TF. 10-Hz Repetitive Transcranial Magnetic Stimulation of the Left Dorsolateral Prefrontal Cortex Reduces Heroin Cue Craving in Long-Term Addicts. Biol Psychiatry. 2016 Aug 1;80(3):e13-4. doi: 10.1016/j.biopsych.2016.02.006. Epub 2016 Feb 12. No abstract available. PMID 26995024
- [Background] Dunlop K, Hanlon CA, Downar J. Noninvasive brain stimulation treatments for addiction and major depression. Ann N Y Acad Sci. 2017 Apr;1394(1):31-54. doi: 10.1111/nyas.12985. Epub 2016 Feb 5. PMID 26849183
- [Background] Carmi L, Tendler A, Bystritsky A, Hollander E, Blumberger DM, Daskalakis J, Ward H, Lapidus K, Goodman W, Casuto L, Feifel D, Barnea-Ygael N, Roth Y, Zangen A, Zohar J. Efficacy and Safety of Deep Transcranial Magnetic Stimulation for Obsessive-Compulsive Disorder: A Prospective Multicenter Randomized Double-Blind Placebo-Controlled Trial. Am J Psychiatry. 2019 Nov 1;176(11):931-938. doi: 10.1176/appi.ajp.2019.18101180. Epub 2019 May 21. PMID 31109199
- [Background] Liu T, Li Y, Shen Y, Liu X, Yuan TF. Gender does not matter: Add-on repetitive transcranial magnetic stimulation treatment for female methamphetamine dependents. Prog Neuropsychopharmacol Biol Psychiatry. 2019 Jun 8;92:70-75. doi: 10.1016/j.pnpbp.2018.12.018. Epub 2018 Dec 31. PMID 30605708
- [Background] Su H, Zhong N, Gan H, Wang J, Han H, Chen T, Li X, Ruan X, Zhu Y, Jiang H, Zhao M. High frequency repetitive transcranial magnetic stimulation of the left dorsolateral prefrontal cortex for methamphetamine use disorders: A randomised clinical trial. Drug Alcohol Depend. 2017 Jun 1;175:84-91. doi: 10.1016/j.drugalcdep.2017.01.037. Epub 2017 Mar 29. PMID 28410525
- [Background] Liu Q, Shen Y, Cao X, Li Y, Chen Y, Yang W, Yuan TF. Either at left or right, both high and low frequency rTMS of dorsolateral prefrontal cortex decreases cue induced craving for methamphetamine. Am J Addict. 2017 Dec;26(8):776-779. doi: 10.1111/ajad.12638. Epub 2017 Nov 14. PMID 29134789